CLINICAL TRIAL: NCT06971003
Title: Community-driven Drug Prevention Implementation Strategies for Native Hawaiian and Pacific Islander Youth in Rural Hawaii
Brief Title: Mohala Na Pua: Community-driven Drug Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Judge Baker Children's Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kelsie Okamura, Implementation Researcher, Judge Baker Children's Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRD003; DP1DA061311 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Adolescent

STUDY DESIGN:
Intervention Model Description: Enrolled students will participate in activities to enhance the implementation of the prevention program in their school. Schools are sequentially recruited each year (i.e., one school will participate per year).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ho'ouna Pono (Experimental): Participants will receive the substance use prevention intervention consisting of (1) a modular classroom curriculum and (2) social media content.
  Interventions: Behavioral: Ho'ouna Pono

INTERVENTIONS:
Behavioral: Ho'ouna Pono — An efficacious culturally grounded substance use prevention intervention developed and tested with Hawaii Island students. Teachers deliver the 11 lesson program through 30-45 minute weekly sessions. The modular intervention can be customized to students by teachers.

SUMMARY:
The goal of this clinical trial is to learn if a substance use prevention intervention decreases substance use, increases resistance skill use, and decreases substance use risk in intermediate school students. The main questions it aims to answer:

Does the intervention decrease 30-day substance use? Does the intervention increase 30-day resistance skill use?

Participants will be asked to participate in the intervention and provide their self-reported answers to behavioral questions before and after the intervention.

DETAILED DESCRIPTION:
Among all ethnic groups in Hawai'i, Native Hawaiian and Pacific Islander youth report the highest rates of substance use, and need for substance use treatment . With the high prevalence of substance use and health disparities among Native Hawaiian, and Pacific Islander (NHPI) communities, research continues to emphasize the need to implement evidence-based prevention programs for youth that are culturally adapted or grounded for indigenous populations. The current five phase, mixed-methods design study aims to use a community-based participatory research approach to implement a culturally grounded, school-based substance use prevention program, Ho'ouna Pono, for NHPI youth across middle/intermediate schools (6th - 8th) in the Windward District of Hawai'i State Department of Education (HIDOE). The current program, Ho'ouna Pono, is a nine-lesson, culturally grounded, video-based, and teacher-delivered substance use prevention curriculum developed on Hawai'i island to build drug resistance skills for middle school students (see Table 3 for specific lesson content). There are three additional modules that are currently being developed. Past program efficacy trials have found statistically significant changes in cigarette/e-cigarette and hard drug use among Native Hawaiian youth on Hawai'i Island, therefore, the research team is interested in evaluating if the intervention will have the same clinical outcome effect with NHPI youth on other islands.

The study focuses on understanding youth substance use and resistance skills prior to and upon completion of the culturally grounded substance use prevention curriculum. The team will be evaluating the program's effects on students' resistance skills development, drug use behaviors, as well as other clinical outcomes data of the intervention, such as drug use behaviors and the utilization of resistance skills.

The overarching research questions are:

* What changes in drug use behaviors are observed among students upon completion of the program?
* What drug resistance strategies did students use upon completion of the program?

ELIGIBILITY:
Inclusion Criteria:

* All students in intermediate schools within the district

Exclusion Criteria:

* None

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
30-day drug use | Through study completion, an average of 10 months
  Self-reported 30-day drug use at baseline and post intervention. Respondents indicate their 30-day behavior in categories including never, only once, a few times, once a week, and almost every day.
30-day prosocial activities | Through study completion, an average of 10 months
  Self-reported 30-day prosocial activities at baseline and post intervention. Respondents indicate their 30-day behavior in categories including never, only once, a few times, once a week, and almost every day.
30-day drug offers | Through study completion, an average of 10 months
  Self-reported 30-day drug offers at baseline and post intervention. Respondents indicate their 30-day behavior in categories including never, only once, a few times, once a week, and almost every day.

SECONDARY OUTCOMES:
30-day resistance skill use | Through study completion, an average of 10 months
  Self-reported resistance skill use to various offers from family and peers at baseline and post intervention. Respondents indicate the extent to which they would use resistance skills in categories including definitely not, probably not, not sure, probably, and definitely. Respondents also indicate how often they have used this response in the last 30 days in categories including never, once, 2-3 times, 4 times, more than 4 times, or not offered.
Risk assessment | Through study completion, an average of 10 months
  Self-reported risk assessment to drug offers at baseline and post intervention. Respondents indicate the extent to which factors might impact their decision in rejecting drug offers in categories including not at all, maybe a little, neutral, a little, a lot.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hawaii State Department of Education - Windward District, Kaneohe, Hawaii
  - The Baker Center for Children and Families, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mohala Na Pua website — https://sites.google.com/view/mohalanapua/home?authuser=0

DOCUMENTS (1):
  • Informed Consent Form (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT06971003/ICF_000.pdf